CLINICAL TRIAL: NCT03666988
Title: A Phase I, Open-label, Dose-escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of GSK3368715 in Participants With Solid Tumors and DLBCL
Brief Title: First Time in Humans (FTIH) Study of GSK3368715 in Participants With Solid Tumors and Diffuse Large B-cell Lymphoma (DLBCL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Overall benefit-risk profile did not support continuation of the study
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 207675; 2018-001629-20 (EudraCT Number)
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Results first posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-02

CONDITIONS: Neoplasms
Keywords: Dose-escalation; First time in humans; Solid tumors; GSK3368715; Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Intervention Model Description: Eligible participants will receive sequential doses of GSK3368715, administered orally once daily in Part 1 of the study and in Part 2, participants will receive RP2D determined in Part 1.
Masking Description: This will be an open-label study. Hence, masking will not be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: GSK3368715 dose escalation (Experimental): Eligible participants with solid relapsed/refractory tumors will receive escalating doses of GSK3368715 at a starting dose of 50 mg, administered orally once daily.
  Interventions: Drug: GSK3368715
- Part 1: GSK3368715 PK/PD/Metabolite/Biomarker (Experimental): Additional participants in Part 1, treated at or close to the expected the maximum tolerated dose (MTD)/RP2D, will be evaluated for metabolic and biomarker profiling. Participants may be enrolled into this cohort(s) even after MTD/RP2D has been identified and Part 2 has been initiated.
  Interventions: Drug: GSK3368715
- Part 1: GSK3368715 Food effect (Experimental): Eligible participants will receive single dose of GSK3368715 at starting dose of 50 mg tablet orally in fasted state followed by fed state in Period 1 and Fed followed by fasted state in Period 2.
  Interventions: Drug: GSK3368715
- Part 2:GSK3368715 dose expansion - DLBCL participants (Experimental): Eligible participants with relapsed/refractory DLBCL will receive RP2D of GSK3368715 established during Part 1, administered orally once daily.
  Interventions: Drug: GSK3368715
- Part 2:GSK3368715 dose expansion-solid tumor participants (Experimental): Eligible participants with relapsed/refractory solid tumors (pancreas cancer, NSCLC, and bladder cancer) will receive RP2D of GSK3368715 established during Part 1, administered orally once daily.
  Interventions: Drug: GSK3368715

INTERVENTIONS:
Drug: GSK3368715 — GSK3368715 will be available with dosing strengths of 25 mg, 100 mg and 250 mg to be administered once daily as an oral capsule.
  Arms: Part 1: GSK3368715 PK/PD/Metabolite/Biomarker; Part 1: GSK3368715 dose escalation; Part 2:GSK3368715 dose expansion - DLBCL participants; Part 2:GSK3368715 dose expansion-solid tumor participants
Drug: GSK3368715 — GSK3368715 will be available in Immediate release (IR) white film coated tablet with dosing strengths of 50 mg, 100 mg and 250 mg to be administered orally once daily .
  Arms: Part 1: GSK3368715 Food effect

SUMMARY:
Arginine methylation mediated by protein arginine methyl-transferases (PRMTs) is an important post-translational modification of proteins involved in a diverse range of cellular processes. Misregulation and overexpression of PRMT1 (a type I PRMT) has been associated with a number of solid and hematopoietic cancers. GSK3368715 leads to inhibition of tumor cell growth across tumor types with cytotoxic response observed in lymphoma, acute myeloid leukemia (AML) and a subset of solid tumor cell lines. This study will assess the safety, pharmacokinetics (PK), pharmacodynamics (PD), food effect and preliminary clinical activity of GSK33368715 in participants with relapsed/refractory DLBCL and selected solid tumors with frequent methyl-thioadenosine phosphorylase (MTAP)-deficiency. The study will consist of two parts. In Part 1 (Dose Escalation) escalating doses of GSK3368715 will be evaluated and recommended phase 2 dose (RP2D) will be established in participants with selected solid relapsed/refractory tumors. Once a RP2D is identified, a food effect sub-study will be initiated to determine the effect of a high-fat, high calorie meal on the bioavailability of GSK3368715. In Part 2 (Dose Expansion), this RP2D will be further investigated in two expansion cohorts; participants with DLBCL (Expansion Cohort 2A) and relapsed/refractory solid tumors including pancreatic, bladder, and non-small cell lung cancer (NSCLC)(Expansion Cohort 2B). The study includes a screening period, an intervention period and follow up.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be >=18 to years of age inclusive, at the time of signing the informed consent.
* Diagnosis of one of the following; Part 1 (Dose Escalation and food effect): Histologically- or cytological-confirmed diagnosis of solid tumor malignancy that is metastatic or non-resectable; have received all standard treatment options or are no longer eligible for additional standard treatment options. Evaluable disease that may be measured directly by the size of the tumor or can be evaluated by other methods. Availability of a biopsy of the tumor tissue obtained at any time from the initial diagnosis to study entry. Although a fresh biopsy, which is obtained during screening, is preferred, archival tumor specimen is acceptable if it is not feasible to obtain a fresh biopsy. For participants in the PK/PD cohort, a fresh biopsy and consent for one on treatment biopsy are required for enrollment. Part 2 (Dose Expansion): Cohort 2A & 2B: The availability of archival tumor tissue, or willingness to undergo a fresh biopsy to determine MTAP status (any archival tumor specimen must have been obtained within 6 months prior to starting study drug unless approved by the study Medical Monitor). Local MTAP or Cyclin Dependent Kinase Inhibitor 2A (CDKN2A) results are acceptable for enrollment, but must be confirmed through central laboratory testing. Cohort 2A: Histologically- or cytological-confirmed diagnosis of DLBCL; relapse or refractory disease after at least 1 but not more than 4 lines of prior therapy; at least 1 measurable site of disease according to the Lugano Classification. The site of disease must be greater than 1.5 centimeter (cm) in the long axis regardless of short axis measurement or greater than 1.0 cm in the short axis regardless of long axis measurement, and clearly measurable in 2 perpendicular dimensions. Cohort 2B: Pancreatic Cancer: Histologically or cytologically confirmed adenocarcinoma of the pancreas; unresectable, locally advanced (Stage III), or metastatic (Stage IV) disease; relapsed or refractory disease after at least 1 prior line of approved, systemic therapy; at least 1 measurable tumor lesion per RECIST 1.1. NSCLC: histologically or cytologically confirmed NSCLC; stage IV disease; tested for presence of echinoderm microtubule-associated protein-like 4- anaplastic lymphoma kinase (EML4-ALK) rearrangement; received at least 2 prior lines of approved, systemic therapy, of which 1 therapy has to be a platinum containing regimen or failed a first-line platinum-containing regimen in combination with an anti- progressive disease (PD1) monocloncal antibody and refused a second-line regimen despite being informed about the different therapeutic options and their specific clinical benefit by the investigator; the content of this informed consent discussion including the therapeutic options reviewed by the investigator need to be documented and the participant needs to sign a specific consent form; at least 1 measurable tumor lesion per RECIST 1.1. Transitional cell carcinoma of the Urothelium: histologically or cytologically confirmed transitional cell carcinoma (TCC) of the urothelium (urinary bladder, urethra, ureter or renal pelvis) including mixed pathology with predominantly (that is [i.e.], > 50 percent of the histopathology sample) TCC with the exception of neuroendocrine or small cell carcinoma; unresectable, locally advanced (T4b) or metastatic (lymph node or visceral) disease; relapsed or refractory disease after at least 1 prior line of approved systemic therapy; at least 1 measurable tumor lesion per RECIST 1.1.
* Adequate organ function as defined by: Absolute neutrophil count (ANC) with a laboratory value of >=1.5 times 10^9 per liter (L); Hemoglobin with a laboratory value of >=9 grams per deciliter (g/dL) for solid malignancy and >=8 g/dL for Non-Hodgkin's lymphoma; Platelets with a laboratory value of >=100 times 10^9/ L; prothrombin time/ International Normalization Ratio (PT/INR) and partial thromboplastin time (PTT) with a laboratory value of <=1.5 times upper limit of normal (ULN), unless participant is receiving systemic anticoagulation (Hematologic); Albumin with a laboratory value of >=2 g/dL, total bilirubin with a laboratory value of <=1.5 times ULN, alanine aminotransferase (ALT) with a laboratory value of <=2.5 times ULN (Part 1 and 2) or <5 times ULN (Part 2 only) is acceptable for participants with documented liver metastases/tumor infiltration (Hepatic); calculated creatinine clearance by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation or measured from 24 h urine with a laboratory value of >= 50 milliliters per min (mL/min) (Renal); Ejection fraction with a laboratory value of >=Lower limit of normal (LLN) by echocardiogram (minimum of 50 percent)/ multigated (radionuclide) angiogram (MUGA), Electrocardiogram (ECG): corrected QT (QTc) interval using Fridericia's formula (QTcF) with a laboratory value of <450 milliseconds (msec) (Cardiac).
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1.
* Able to swallow and retain orally-administered medication.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies; is not a woman of childbearing potential (WOCBP) or is a WOCBP and using a contraceptive method that is highly effective, with a failure rate of <1 percent, during the intervention period and for at least 120 days, corresponding to the time needed to eliminate any study intervention(s) (example given [e.g.], 5 terminal half-lives) after the last dose of study intervention. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. A WOCBP must have a negative highly sensitive pregnancy test (urine as required by local regulations) within 7 days before the first dose of study intervention. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy. Male participants are eligible to participate if they agree to the following during the intervention period and for at least 100 days, corresponding to time needed to eliminate study intervention(s) (e.g., 5 terminal half-lives) plus 90 days after the last dose of study intervention: Refrain from donating sperm plus either: Be abstinent from heterosexual or homosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or must agree to use contraception/barrier as detailed below; agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant; agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History of malignancy other than the disease under study. Participants who have been disease-free for 5 years, or participants with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible. Participants with second malignancies that are indolent or definitively treated may be enrolled even if less than 5 years have elapsed since treatment.
* Primary central nervous system (CNS) tumors, Glioblastoma multiforme (GBM), symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. Participants previously treated for these conditions that have had stable CNS disease (verified with consecutive imaging studies) for >1 months, are asymptomatic and off corticosteroids, or are on stable dose of corticosteroids for at least 1 month prior to study Day 1 are permitted. Stability of brain metastases must be confirmed with imaging. Participants treated with gamma knife therapy can be enrolled 2 weeks post-procedure as long as there are no post-procedure complications/they are stable.
* Any severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, cardiac disease, or clinically significant bleeding episodes, or active infection).
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator.
* Any clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels.
* History of known human immunodeficiency virus (HIV) infection or positive HIV test result at screening.
* Presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening to first dose of study intervention.
* Any of the following cardiac abnormalities: Uncontrolled high blood pressure; any history of coronary artery disease, including acute coronary syndromes, myocardial infarction, unstable angina, and history of coronary angioplasty, or stenting; presence of a cardiac pacemaker or implanted defibrillator; atrioventricular (AV)-block (asymptomatic 2nd degree Type II or 3rd degree and any degree AV block if related to heart disease or if symptomatic), right bundle branch block (RBBB), left bundle branch block (LBBB), and any fasicular hemiblocks; A QRS interval at Screening or Baseline >110 msec; participants with any symptomatic or sustained arrhythmias (past or present), including but not limited to: Atrial fibrillation, Atrial flutter, Ventricular tachycardia, Ventricular fibrillation, Supraventricular tachycardia; Current or past congestive heart failure; Evidence of a left ventricular ejection fraction below the institutional lower limit of normal on Screening echocardiogram; Evidence of significant structural heart disease on echocardiography at Screening (including any valvular disease greater than "mild" in severity); Cardiac troponin > upper limit of the reference range at Screening.
* Treatment with any local or systemic anti-neoplastic therapy or investigational anticancer agent within 14 days or 4 half-lives, whichever is longer, up to a maximum wash-out period of 28 days prior to initiation of study drug administration. Anti-androgen therapies for prostate cancer, such as bicalutamide, must be stopped 28 days prior to first dose of GSK3368715. Second-line hormone therapies such as enzalutamide or abiraterone should be stopped 14 days prior to enrolment. Participants with prostate cancer may remain on luteinizing hormone-releasing hormone (LHRH) agonists or antagonists and/or low-dose prednisone or prednisolone (up to 10 milligrams per day [mg/day]). Nitrosureas and mitomycin C must be stopped within 42 days prior to first dose of GSK3368715.
* Allogeneic hematopoietic stem-cell transplantation.
* Toxicities from previous anti-cancer therapies have not resolved to Baseline or National Cancer Institute (NCI) CTCAE V5.0. <=Grade 1 (except fatigue and alopecia [permissible at any grade] and peripheral neuropathy [which must be <= Grade 2]) at the time of starting study intervention.
* Major surgery (i.e. requiring general anesthesia) within 3 weeks before screening, or not fully recovered from major surgery, or major surgery planned during study participation. Planned surgical procedures to be conducted under local anesthesia are allowed.
* Prior organ transplantation.
* Concurrent anti-coagulation therapy. Treatment with low-molecular heparin is allowed.
* Current use of a prohibited medication or planned use of any forbidden medications during intervention with GSK3368715.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Participant is considered high-risk for VTE as defined by either Khorana Score of greater than or equal to 3 or prior medical history of VTE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (5):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
- GSK Investigational Site, Melbourne, Victoria, Australia
- GSK Investigational Site, Toronto, Ontario, Canada
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] El-Khoueiry AB, Clarke J, Neff T, Crossman T, Ratia N, Rathi C, Noto P, Tarkar A, Garrido-Laguna I, Calvo E, Rodon J, Tran B, O'Dwyer PJ, Cuker A, Abdul Razak AR. Phase 1 study of GSK3368715, a type I PRMT inhibitor, in patients with advanced solid tumors. Br J Cancer. 2023 Aug;129(2):309-317. doi: 10.1038/s41416-023-02276-0. Epub 2023 May 26. PMID 37237172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was planned as a 2-part, first time in human study in participants with solid tumors and Diffuse Large B-Cell Lymphoma (DLBCL). Part 1 was planned to include dose escalation and food effect cohorts and Part 2 was an expansion cohort.
Pre-assignment Details: This study was terminated early during Part 1 as the benefit/risk assessment did not favor continuation of the study and therefore, Part 1: Food effect cohorts and Part 2 were not conducted. Total 31 participants were enrolled in Part 1 of the study.
Groups:
- Part 1 GSK3368715 50mg: Participants with solid relapsed/refractory tumors were administered once daily oral dose of GSK3368715 50 milligrams (mg).
- Part 1 GSK3368715 100mg: Participants with solid relapsed/refractory tumors were administered once daily oral dose of GSK3368715 100mg.
- Part 1 GSK3368715 200mg: Participants with solid relapsed/refractory tumors were administered once daily oral dose of GSK3368715 200mg.
- Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed: Participants with solid relapsed/refractory tumors were planned to receive once daily oral dose of GSK3368715 with a tablet formulation in the fasted state followed by fed state at or near the recommended Phase II dose (RP2D).
- Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted: Participants with solid relapsed/refractory tumors were planned to receive once daily oral dose of GSK3368715 with a tablet formulation in the fed state followed by fasted state at or near the RP2D.
- Part 2 GSK3368715 Expansion Cohort: Participants with DLBCL were planned to receive recommended Phase II dose (RP2D) based on Part 1 data.
Period: Part 1 (Up to 28 Months)
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted | Part 2 GSK3368715 Expansion Cohort
Started | 3 | 16 | 12 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 16 | 12 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 3 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Disease Progression | 2 | 14 | 7 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Up to 48 Months)
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted | Part 2 GSK3368715 Expansion Cohort
Started | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated early during Part 1 as the benefit/risk assessment did not favor continuation of the study, therefore Part 1: Food effect cohorts and Part 2 were not conducted.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted | Part 2 GSK3368715 Expansion Cohort | Total
Number analyzed (Participants) | 3 | 16 | 12 | 0 | 0 | 0 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] — Study was terminated early during Part 1 as the benefit/risk assessment did not favor continuation of the study, therefore Part 1: Food effect cohorts and Part 2 were not conducted.
  Years | 68.0 (6.56) | 55.5 (15.12) | 59.7 (10.89) |  |  |  | 58.3 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants] — Study was terminated early during Part 1 as the benefit/risk assessment did not favor continuation of the study, therefore Part 1: Food effect cohorts and Part 2 were not conducted.
  Participants
    Female | 2 | 4 | 3 | 0 | 0 | 0 | 9
    Male | 1 | 12 | 9 | 0 | 0 | 0 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Study was terminated early during Part 1 as the benefit/risk assessment did not favor continuation of the study, therefore Part 1: Food effect cohorts and Part 2 were not conducted.
  Participants
    Asian - East Asian Heritage | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Asian - South East Asian Heritage | 0 | 1 | 1 | 0 | 0 | 0 | 2
    White - Arabic/North African Heritage | 0 | 2 | 4 | 0 | 0 | 0 | 6
    White - White/Caucasian/European Heritage | 3 | 12 | 6 | 0 | 0 | 0 | 21
    Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT is considered by the investigator to be clinically relevant,attributed event during the first 21days of intervention meeting the following criteria:Non-hematologic toxicity:Aspartate Aminotransferase(AST)/Alanine Aminotransferase(ALT) Grade 3/4,ALT>=5 times Upper limit of Normal(ULN),ALT>=3times ULN(>=4 weeks),ALT>=3 times ULN plus(+)bilirubin>=2 times ULN,ALT >= 3 times ULN+liver symptoms or International Normalization Ratio(INR)>1.5.Nausea:Grade 3;Vomiting or diarrhea:Grade3/4(>3days);Fatigue:Grade 3(>5days).Hypertension:Uncontrolled Grade 3/4.Electrocardiogram(ECG)-change:>20 milliseconds(msec) QRS extension.Lab abnormality:uncontrolled Grade3(>3days)/Grade4.Hematologic toxicity:Neutropenia:uncontrolled Grade3(>3days)/febrile neutropenia/Grade 4.Thrombocytopenia:uncontrolled Grade 3(>3days)/Grade 3(clinically significant Hemorrhage)/Grade 4.Venous thromboembolism (VTE):Grade2 needing systemic anticoagulation/Grade>=3 during the first 8 weeks or if sooner,study discontinuation
Time Frame: Up to 21 days
Population: All-Treated Population included all participants who received at least one dose of GSK3368715. Data was not collected for Part 1: Food Effect Cohorts, as the study was terminated early during Part 1 and hence no participants were enrolled in Part 1: Food Effect Cohorts
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Food Effect Cohort: GSK3368715 Fasted Followed by Fed: Participants with solid relapsed/refractory tumors were planned to receive once daily oral dose of GSK3368715 with a tablet formulation in the fasted state followed by fed state at or near the recommended Phase II dose (RP2D).
- Part 1: Food Effect Cohort: GSK3368715 Fed Followed by Fasted: Participants with solid relapsed/refractory tumors were planned to receive once daily oral dose of GSK3368715 with a tablet formulation in the fed state followed by fasted state at or near the RP2D.
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg | Part 1: Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1: Food Effect Cohort: GSK3368715 Fed Followed by Fasted
Number analyzed (Participants) | 3 | 16 | 12 | 0 | 0
Participants | 0 | 0 | 3 |  |

2. Primary Outcome: Part 1: Number of Participants With Non-Serious Adverse Events (Non-SAEs) and SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Any untoward event resulting in death, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment is categorized as SAE.
Time Frame: Up to 28 months
Population: All-Treated Population. Data was not collected for Part 1: Food Effect Cohorts, as the study was terminated early during Part 1 and hence no participants were enrolled in Part 1: Food Effect Cohorts
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted
Number analyzed (Participants) | 3 | 16 | 12 | 0 | 0
Participants
  Any Non-SAE | 3 | 15 | 9 |  |
  Any SAE | 2 | 4 | 6 |  |

3. Primary Outcome: Part 1: Number of Participants With AEs by Severity Grades
Description: All adverse events were analyzed using National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0. Graded from Grade 1: mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL), Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL, Grade 4: Life-threatening consequences; urgent intervention indicated, Grade 5: death related AE. Higher grade indicates more severe condition. Number of participants with maximum severity grades are presented.
Time Frame: Up to 28 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted
Number analyzed (Participants) | 3 | 16 | 12 | 0 | 0
Participants
  Grade 1 | 1 | 0 | 2 |  |
  Grade 2 | 1 | 9 | 1 |  |
  Grade 3 | 1 | 5 | 5 |  |
  Grade 4 | 0 | 1 | 2 |  |
  Grade 5 | 0 | 0 | 2 |  |

4. Primary Outcome: Part 2: Percentage of Participants Achieving Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a confirmed complete response (CR) or a partial response (PR). Participants with solid tumor were planned to be assessed per Response Criteria for Solid Tumors (RECIST) 1.1 and DLBCL participants were planned to be assessed per Lugano Criteria. This analysis was planned but not performed for Part 2 as the study was terminated during Part 1.
Time Frame: Up to 48 months
Population: All-Treated Population. Data was not collected in Part 2 as the study was terminated early during Part 1 and hence no participant was enrolled in Part 2.
Arm/Group | Part 2 GSK3368715 Expansion Cohort
Number analyzed (Participants) | 0

5. Secondary Outcome: Part 1: Percentage of Participants Achieving Best Overall Response Rate
Description: Overall response rate is defined as the percentage of participants with a confirmed complete response (CR) or a partial response (PR). Participants with solid tumor were assessed per Response Criteria for Solid Tumors (RECIST) 1.1 and DLBCL participants were assessed per Lugano Criteria. The best ORR was recorded from the start of the intervention until disease progression/recurrence and was determined based on the investigator's assessment of response at each time point. The percentage of participants achieving best overall response rate have been presented.
Time Frame: Up to 28 months
Population: All Treated Population. Data was not collected for Part 1: Food Effect Cohorts, as the study was terminated early during Part 1 and hence no participants were enrolled in Part 1: Food Effect Cohorts
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted
Number analyzed (Participants) | 3 | 16 | 12 | 0 | 0
Percentage of participants | 0 | 0 | 0 |  |

6. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) Following Administration of GSK3368715
Description: Blood samples were collected at indicated time points. The pharmacokinetic (PK) parameters were calculated by non-compartmental analysis. PK Population included all participants in the All-Treated population from whom at least one PK sample was obtained, analyzed, and was measurable.
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2 ,3 ,4 ,6, 8, 12, 24, 48, 72 hours post-dose on Day 1; Pre-dose,30 minutes, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 15
Population: PK Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). Data was not collected for Part 1: Food Effect Cohorts, as the study was terminated early during Part 1 and hence no participants were enrolled in Part 1: Food Effect Cohorts
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg
Number analyzed (Participants) | 3 | 16 | 12
Nanograms per milliliter
  GSK3368715 Day 1,n=3,16,12 | 107.166 (48.81) | 197.420 (112.05) | 336.771 (72.57)
  GSK3368715 Day 15,n=3,14,9: number analyzed (Participants) | 3 | 14 | 9
  GSK3368715 Day 15,n=3,14,9 | 111.898 (48.51) | 375.485 (79.86) | 729.196 (42.82)

7. Secondary Outcome: Part 1: Time to Reach Cmax (Tmax) Following Administration of GSK3368715
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on Day 1; Pre-dose,30 minutes, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 15
Population: PK Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).Data was not collected for Part 1: Food Effect Cohorts, as the study was terminated early during Part 1 and hence no participants were enrolled in Part 1: Food Effect Cohorts
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg
Number analyzed (Participants) | 3 | 16 | 12
Hours
  GSK3368715 Day 1,n=3,16,12 | 0.5326 (180.404) | 0.6821 (94.273) | 1.1594 (86.483)
  GSK3368715 Day 15,n=3,14,9: number analyzed (Participants) | 3 | 14 | 9
  GSK3368715 Day 15,n=3,14,9 | 1.7023 (132.169) | 0.8080 (44.215) | 0.9946 (66.296)

8. Secondary Outcome: Part 1: Area Under the Concentration Time Curve From Time Zero to Last Time of Quantifiable Concentration (AUC [0-t]) Following Administration of GSK3368715
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg
Number analyzed (Participants) | 3 | 16 | 12
Hour*nanogram per milliliter
  GSK3368715 Day 1,n=3,16,12 | 283.4828 (32.756) | 483.1405 (107.980) | 1400.0804 (64.718)
  GSK3368715 Day 15,n=3,14,9: number analyzed (Participants) | 3 | 14 | 9
  GSK3368715 Day 15,n=3,14,9 | 437.2790 (91.371) | 1569.2088 (64.014) | 4870.1952 (45.623)

9. Secondary Outcome: Part 1: AUC From Time Zero Extrapolated to Infinite Time (AUC [0-infinity]) Following Administration of GSK3368715
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on Day 1
Population: PK Population.Only those participants (par) with data available at specified data points were analyzed.Data not collected for Part (P)1:Food Effect Cohorts (FEC),as study was terminated early during P1;hence no par were enrolled in P1:FEC.AUC(0-infinity) could not be calculated for par in "P1 GSK3368715 50mg" arm,as atleast 3 data points are required in terminal elimination phase within same par;this criteria could not be fulfilled due to insufficient data above limit of quantification
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg
Number analyzed (Participants) | 0 | 2 | 4
Hour*nanogram per milliliter |  | 1217.5147 (27.619) | 1674.8304 (50.515)

10. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero to the Predose of the Next Dose [AUC (0-tau)] Following Administration of GSK3368715
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 30 minutes, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 15
Population: PK Population. Only those participants with data available at the specified data points were analyzed. Data was not collected for Part 1: Food Effect Cohorts, as the study was terminated early during Part 1 and hence no participants were enrolled in Part 1: Food Effect Cohorts
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg
Number analyzed (Participants) | 2 | 14 | 9
Hour*nanogram per milliliter | 581.9071 (101.434) | 1573.8450 (64.183) | 4861.3917 (45.288)

11. Secondary Outcome: Part 1: Trough (Pre-dose) Concentration (Ctau) Following Administration of GSK3368715
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis. Not applicable (NA) indicates that data could not be calculated as these were derivate values which were below the lower limit of quantification.
Time Frame: Pre-dose on Day 1 and Day 15
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg
Number analyzed (Participants) | 3 | 16 | 11
Nanogram per milliliter
  GSK3368715 Day 1,n=3,16,11 | 5.150 (NA) — Data could not be calculated as these were derivate values which were below the lower limit of quantification. | 7.880 (18.46) | 12.642 (73.85)
  GSK3368715 Day 15,n=3,14,10: number analyzed (Participants) | 3 | 14 | 10
  GSK3368715 Day 15,n=3,14,10 | 13.609 (120.74) | 26.421 (69.92) | 89.383 (70.43)

12. Secondary Outcome: Part 1: Time Invariance Ratio Following Administration of GSK3368715
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis. Time invariance was calculated as the ratio of AUC(0-24) on Day 15 / AUC (0-infinity) on Day 1 for GSK3368715.
Time Frame: Pre-dose, 15, 30 minutes, 1 ,1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on Day 1; Pre-dose, 30 minutes,1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 15
Population: PK Population. Only those participants with data available at the specified data points were analyzed. Data was not collected for Part 1: Food Effect Cohorts, as the study was terminated early during Part 1 and hence no participants were enrolled in Part 1: Food Effect Cohorts. Time invariance computation is dependent on AUC(0-infinity) and since AUC(0-infinity) could not be computed for participants in "Part 1 GSK3368715 50mg" arm, time invariance was not computable as well.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg
Number analyzed (Participants) | 0 | 2 | 4
Ratio |  | 1.6007 (15.614) | 2.9492 (43.451)

13. Secondary Outcome: Part 1: Accumulation Ratio Following Administration of GSK3368715
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis. Accumulation ratio (AR) was calculated as the ratio of AUC(0-24) on Day 15/Day 1 for GSK3368715.
Time Frame: Pre-dose, 15, 30 minutes, 1 ,1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on Day 1; Pre-dose, 30 minutes, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 15
Population: PK Population.Only those participants with data available at the specified data points were analyzed. Data was not collected for Part 1: Food Effect Cohorts,as study was terminated early during Part 1 and hence no participants were enrolled in Part 1: Food Effect Cohorts. Accumulation ratio could not be derived for "Part 1 GSK3368715 50mg" arm because there were no participant with AUC(0-24) values at both Day 1 and Day 15; hence, paired results were not available to calculate Accumulation ratio
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg
Number analyzed (Participants) | 0 | 7 | 9
Ratio |  | 2.6276 (37.761) | 3.5953 (40.900)

14. Secondary Outcome: Part 1: Food Effect Cohorts: Cmax Following Administration of GSK3368715
Description: Blood samples were planned to be collected at indicated time points in food effect cohorts (fasted followed by fed state and fed followed by fasted state). Samples were not collected due to early termination of study during Part 1; therefore, no analysis could be performed.
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on Day 1; Pre-dose, 1 and 4 hours post dose on Day 8, Pre-dose, 30 minutes, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 15
Population: PK Population. Data was not collected for Part 1: Food Effect Cohorts, as the study was terminated early during Part 1 and hence no participants were enrolled in Part 1: Food Effect Cohorts
Arm/Group | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Part 1: Food Effect Cohorts: Tmax Following Administration of GSK3368715
Description: Blood samples were planned to be collected at indicated time points in food effect cohorts (fasted followed by fed state and fed followed by fasted state). Samples were not collected due to early termination of the study during Part 1; therefore, no analysis could be performed.
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on Day 1; Pre-dose, 1 and 4 hours post dose on Day 8, Pre-dose, 30 minutes, 1 ,2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 15
Population: as for outcome 14
Arm/Group | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Part 1: Food Effect Cohorts: AUC (0-t) Following Administration of GSK3368715
Description: as for outcome 15
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on Day 1; Pre-dose, 1 and 4 hours post dose on Day 8, Pre-dose,30 minutes, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 15
Population: as for outcome 14
Arm/Group | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Part 1: Food Effect Cohorts: AUC (0-infinity) Following Administration of GSK3368715
Description: as for outcome 15
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on Day 1; Pre-dose, 1 and 4 hours post dose on Day 8, Pre-dose,30 minutes,1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 15
Population: as for outcome 14
Arm/Group | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Part 1: Food Effect Cohorts: AUC (0-tau) Following Administration of GSK3368715
Description: as for outcome 15
Time Frame: as for outcome 14
Population: as for outcome 14
Arm/Group | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Part 2: Number of Participants With Non-SAEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Any untoward event resulting in death, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment is categorized as serious adverse event (SAE). This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 48 months
Population: All Treated Population. Data was not collected as the study was terminated early during Part 1 and hence no participants were enrolled in Part 2.
Arm/Group | Part 2 GSK3368715 Expansion Cohort
Number analyzed (Participants) | 0

20. Secondary Outcome: Part 2: Number of Participants With AEs by Severity Grades
Description: All adverse events were analyzed using National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0. Graded from Grade 1: mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL), Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL, Grade 4: Life-threatening consequences; urgent intervention indicated, Grade 5: death related AE. Higher grade indicates more severe condition. Number of participants with maximum severity grades were presented. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 48 months
Population: as for outcome 19
Arm/Group | Part 2 GSK3368715 Expansion Cohort
Number analyzed (Participants) | 0

21. Secondary Outcome: Part 2: Progression-free Survival (PFS)
Description: PFS is defined as the time from the first dose of study intervention to disease progression or death due to any cause, whichever occurs earlier. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 48 months
Population: as for outcome 19
Arm/Group | Part 2 GSK3368715 Expansion Cohort
Number analyzed (Participants) | 0

22. Secondary Outcome: Part 2: Cmax Following Administration of GSK3368715
Description: Blood samples were planned to be collected for PK analysis of GSK3368715. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5 ,2 ,3 ,4 ,6, 8, 12, 24, 48, 72 hours post-dose on Day 1; Pre-dose,30 minutes, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 15
Population: PK Population. Data was not collected as the study was terminated early during Part 1 and hence no participants were enrolled in Part 2.
Arm/Group | Part 2 GSK3368715 Expansion Cohort
Number analyzed (Participants) | 0

23. Secondary Outcome: Part 2: Tmax Following Administration of GSK3368715
Description: as for outcome 22
Time Frame: as for outcome 7
Population: as for outcome 22
Arm/Group | Part 2 GSK3368715 Expansion Cohort
Number analyzed (Participants) | 0

24. Secondary Outcome: Part 2: AUC (0-t) Following Administration of GSK3368715
Description: as for outcome 22
Time Frame: as for outcome 7
Population: as for outcome 22
Arm/Group | Part 2 GSK3368715 Expansion Cohort
Number analyzed (Participants) | 0

25. Secondary Outcome: Part 2: AUC (0-infinity) Following Administration of GSK3368715
Description: Blood samples were planned to be collected for PK analysis of GSK3368715 . This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Pre-dose, 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on Day 1
Population: as for outcome 22
Arm/Group | Part 2 GSK3368715 Expansion Cohort
Number analyzed (Participants) | 0

26. Secondary Outcome: Part 2: AUC (0-tau) Following Administration of GSK3368715
Description: as for outcome 22
Time Frame: Pre-dose, 30 minutes, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 15
Population: as for outcome 22
Arm/Group | Part 2 GSK3368715 Expansion Cohort
Number analyzed (Participants) | 0

27. Secondary Outcome: Part 2: Ctau Following Administration of GSK3368715
Description: Blood samples were planned to be collected for pharmacokinetic analysis of GSK3368715. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Pre-dose on Day 1 and Day 15
Population: as for outcome 22
Arm/Group | Part 2 GSK3368715 Expansion Cohort
Number analyzed (Participants) | 0

28. Secondary Outcome: Part 2: Time Invariance Ratio Following Administration of GSK3368715
Description: as for outcome 27
Time Frame: as for outcome 12
Population: as for outcome 22
Arm/Group | Part 2 GSK3368715 Expansion Cohort
Number analyzed (Participants) | 0

29. Secondary Outcome: Part 2: Accumulation Ratio Following Administration of GSK3368715
Description: as for outcome 22
Time Frame: as for outcome 13
Population: as for outcome 22
Arm/Group | Part 2 GSK3368715 Expansion Cohort
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-serious adverse events (Non-SAEs) were collected from the start of the study treatment up to 28 months in Part 1.
Description: All Treated Population included all participants who received at least one dose of GSK3368715. Study was terminated early during Part 1 as the benefit/risk assessment did not favor continuation of the study; therefore, Part 1: Food effect cohorts and Part 2 were not conducted.
Arm/Group | Part 1 GSK3368715 50mg | Part 1 GSK3368715 100mg | Part 1 GSK3368715 200mg | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted | Part 2 GSK3368715 Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/16 | 0/12 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/16 | 6/12 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 15/16 | 9/12 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 GSK3368715 50mg (N=3) | Part 1 GSK3368715 100mg (N=16) | Part 1 GSK3368715 200mg (N=12) | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed (N=0) | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted (N=0) | Part 2 GSK3368715 Expansion Cohort (N=0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 GSK3368715 50mg (N=3) | Part 1 GSK3368715 100mg (N=16) | Part 1 GSK3368715 200mg (N=12) | Part 1:Food Effect Cohort: GSK3368715 Fasted Followed by Fed (N=0) | Part 1:Food Effect Cohort: GSK3368715 Fed Followed by Fasted (N=0) | Part 2 GSK3368715 Expansion Cohort (N=0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (6) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 6 (11) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03666988/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03666988/SAP_001.pdf